CLINICAL TRIAL: NCT02299609
Title: Therapeutic Effect of Ultrasound Beams as an Adjunct to Reperfusion Therapy in STEMI
Brief Title: Ultrasound Beams as an Adjunct to Reperfusion Therapy in STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Ramazan Akdemir, Prof. Ramazan Akdemir, MD, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CCTSAU1400
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Myocardial Infarction; ST Elevation Myocardial Infarction
Keywords: C14.280.647.500
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beam Receiver (Active Comparator): Philips HD11 XE® 30 min qid x 4 days
  Interventions: Other: Ultrasound beams Philips HD11 XE®
- Beam Non-Receiver (Sham Comparator): Philips HD11 XE® (ultrasound turned-off) 30 min qid x 4 days
  Interventions: Other: Ultrasound beams Philips HD11 XE®

INTERVENTIONS:
Other: Ultrasound beams Philips HD11 XE® — Ultrasound beams used during standard echocardiography

SUMMARY:
Successfully perfused STEMI patients will receive routine transthoracic echocardiography qid for 4 days or placebo. Myocardial function and infarct size will be evaluated at 3 and 6 months.

DETAILED DESCRIPTION:
Patients who had acute STEMI and successfully reperfused by either thrombolytic therapy or primary angioplasty and stenting will be included this study.

A basal routine echocardiography will be obtained in all patients after reperfusion therapy. Thereafter, patients will be divided into two groups: 1.Treatment group will receive transthoracic echocardiography using Philips HD11 XE ® for 30 minutes qid for 4 days. 2. Placebo group will have the same Philips HD11 XE ® echo transducer applied for the same time and duration on their chest but with the ultrasound turned-off. Detailed left and right ventricle function as well as performance index and stress-strain imaging will be obtained and analyzed at 3 and 6 months.

ELIGIBILITY:
Inclusion criteria:

-Patients presenting within 12 hours of their first ST- elevation myocardial infarction that is successfully reperfused; and completed baseline echocardiographic evaluation and accepted participation in the study

Exclusion criteria:

Patients:

* With prior ST- elevation myocardial infarction
* Patients presenting >12hrs
* Not successfully reperfused
* Not completed baseline ECHO evaluation,
* Not accepting participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Increase in left ventricular function | At 3 and 6 months
  Ultrasound beams during echocardiography application expected to ameliorate the left ventricle function

SECONDARY OUTCOMES:
Decrease in infarct size | At 3 and 6 months
  Ultrasound beams during echocardiography application expected to decrease infarct size

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Akdemir, MD, Study Chair — Sakarya University
Locations (1):
- Sakarya University, Faculty of Medicine, Sakarya, Turkey (Türkiye)

REFERENCES:
- [Result] Ling ZY, Shu SY, Zhong SG, Luo J, Su L, Liu ZZ, Lan XB, Yuan GB, Zheng YY, Ran HT, Wang ZG, Yin YH. Ultrasound targeted microbubble destruction promotes angiogenesis and heart function by inducing myocardial microenvironment change. Ultrasound Med Biol. 2013 Nov;39(11):2001-10. doi: 10.1016/j.ultrasmedbio.2013.06.003. Epub 2013 Aug 19. PMID 23969167
- [Result] Nazer B, Gerstenfeld EP, Hata A, Crum LA, Matula TJ. Cardiovascular applications of therapeutic ultrasound. J Interv Card Electrophysiol. 2014 Apr;39(3):287-94. doi: 10.1007/s10840-013-9845-z. Epub 2013 Dec 3. PMID 24297498